CLINICAL TRIAL: NCT04738175
Title: A Randomized, Controlled Study to Evaluate the Safety and Efficacy of a Single Dose of STI-2020 (COVI-AMG™) to Treat COVID-19
Brief Title: Study to Evaluate the Safety and Efficacy of a Single Dose of STI-2020 (COVI-AMG™) to Treat COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A different study will be conducted.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMG-COV-201-BR
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-AMG (Experimental): 40 mg, 100 mg, or 200 mg of COVI-AMG will be administered
  Interventions: Biological: COVI-AMG
- Placebo (Placebo Comparator): Placebo will be administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-AMG — COVI-AMG is a fully human SARS-CoV-2 neutralizing monoclonal antibody (mAb)
  Other Names: STI-2020
  Arms: COVI-AMG
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
Subjects will receive a single injection of 40, 100, or 200 mg COVI-AMG or placebo via IV push.

DETAILED DESCRIPTION:
Subjects will receive a single injection of 40, 100, or 200 mg COVI-AMG or placebo via IV push. Subjects will be followed for 70 days after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with recent COVID-19 diagnosis with mild or moderate symptoms lasting less than 7 days prior to Screening and not requiring imminent hospitalization
* No medical or psychiatric conditions that could put the subject at risk
* Willing to follow contraception guidelines

Exclusion Criteria:

* Clinical signs of COVID-19 indicative of impending hospitalization
* Documented infection in addition to COVID-19 that requires systemic treatment
* Medical condition that could adversely impact safety, in the Investigator's opinion
* Is or planning to be pregnant or lactating
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies (mAbs) against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit
* Has received or will receive during study participation a vaccine for COVID-19
* Has participated in clinical trial protocols in the last 12 months, unless the Investigator believes that there may be a direct benefit to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events by type, frequency, severity, and causality (safety) | Randomization through study completion at Day 70
  Safety as assessed by incidence of adverse events by type, frequency, severity, and causality
Changes in viral shedding from Baseline to Day 15 | Randomization to Day 15
  Changes in viral shedding from Baseline to Day 15

SECONDARY OUTCOMES:
Changes in viral shedding from Baseline to Day 8, 29, 43, and 70 | Randomization to Day 8, 29, 43, 70
  Changes in viral shedding from Baseline to Day 8, 29, 43, and 70
Time to viral RNA negativity | Randomization through study completion at Day 70
  Time to viral RNA negativity using nasopharyngeal reverse transcription PCR
Time to resolution of symptoms | Randomization through study completion at Day 70
  Time to resolution of symptoms as assessed by the COVID-19 PRO instrument

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics